CLINICAL TRIAL: NCT05208138
Title: Feasibility and Safety of Robotic Bariatric Surgery Using the SenhanceTM Surgical System: a Pilot Study
Brief Title: Feasibility and Safety of Robotic Bariatric Surgery Using the SenhanceTM Surgical System
Acronym: RoboBar
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: leasing of the Senhance system ended
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STD0005853
Record Dates: First submitted 2021-12-27; First posted 2022-01-26 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Bariatric Surgery Candidate
Keywords: Bariatric Surgery; Robotic Surgery

STUDY DESIGN:
Intervention Model Description: Prospective single arm, two-stage phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Bariatric operation with the Senhance surgical system
  Interventions: Device: Senhance Surgical System from Asensus

INTERVENTIONS:
Device: Senhance Surgical System from Asensus — Bariatric operation with the Senhance Surgical System

SUMMARY:
Evaluating feasibility and safety of the Senhance Surgical System with digital laparoscopy in bariatric surgery.

DETAILED DESCRIPTION:
The introduction of laparoscopy in bariatric surgery is considered a milestone to improve postoperative outcomes in terms of less complications and shorter hospital stay. Furthermore, conversion into open surgery is associated with higher postoperative morbidity and mortality in bariatric surgery. Nevertheless, the laparoscopic technique has several drawbacks as lack of tactile feedback, limited degrees of freedom of the laparoscopic instruments, bad depth perception and limited field of view and therefore a flat learning curve.

Senhance Surgical System from Asensus Surgical is an innovative robotic technique which presents haptic feedback, an eyetracker system, microinvasive surgery (with 3mm instruments), reusable instruments and a lower docking time when compared to usual robotic systems.

The use of this new technology has not been systematically analysed in bariatric surgery. Nevertheless, its use is expected to be safe and efficient and may also present some advantages over conventional laparoscopic surgery.

The primary endpoint of the study is the safety of this new robotic platform in bariatric surgery (intraoperative complications, postoperative morbidity, and postoperative mortality). Secondary outcome is the feasibility of this new technology in bariatric surgery (docking time, operation time, conversion rate, length of hospital stay, and rehospitalisation rate).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* ≥ 18 years old
* Capable of judgment
* Patient eligible for laparoscopic bariatric surgery according to the SMOB (Swiss Study Group for Morbid Obesity) -Criteria and having a bariatric operation (including Sleeve gastrectomy, Y-Roux gastric bypass, Omega-loop gastric bypass) using SenhanceTM Surgical System

Exclusion Criteria:

* < 18 years of age
* Participants incapable of judgment or participants under tutelage
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* No informed consent signed
* Women who are pregnant
* High risk patients (immunosuppression, myopathy, liver cirrhosis, severe heart or lung disease, renal failure)
* Contra-indication for laparoscopic surgery
* Prior upper gastro intestinal tract operations (such as hepatobiliary, pancreatic, gastrooesophageal, anti-reflux, bariatric surgery or splenectomy except cholecystectomy) or open surgery with incision above the umbilicus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Rate of intraoperative bleeding using the Senhance Surgical System in bariatric surgery | During operation, up to 2 hours
  Number of patients with intraoperative bleeding
Rate of intraoperative organ lesion using the Senhance Surgical System in bariatric surgery | During operation, up to 2 hours
  Number of patients with intraoperative organ lesion
Rate of procedure interruption using the Senhance Surgical System in bariatric surgery | During operation, up to 2 hours
  Number of patients with procedure interruption
Rate of postoperative bleeding using the Senhance Surgical System in bariatric surgery | up to 30 days postoperatively
  Number of patients with postoperative bleeding
Rate of anastomotic or staple line leakage using the Senhance Surgical System in bariatric surgery | up to 30 days postoperatively
  Number of patients with anastomotic or staple line leakage
Rate of surgical site infection using the Senhance Surgical System in bariatric surgery | up to 30 days postoperatively
  Number of patients with surgical site infection (deep or superficial)
Rate of cardiovascular complication using the Senhance Surgical System in bariatric surgery | up to 30 days postoperatively
  Number of patients with a cardiovascular complication
Rate of respiratory complication using theSenhance Surgical System in bariatric surgery | up to 30 days postoperatively
  Number of patients with a respiratory complication
Rate of thromboembolic complication using the Senhance Surgical System in bariatric surgery | up to 30 days postoperatively
  Number of patients with a thromboembolic complication
Rate of renal complication using the Senhance Surgical System in bariatric surgery | up to 30 days postoperatively
  Number of patients with a renal complication

SECONDARY OUTCOMES:
Feasibility of the Senhance Surgical System in bariatric surgery | During operation, up to 2 hours
  Operation time
Feasibility of the Senhance Surgical System in bariatric surgery | During operation, up to 2 hours
  Docking time
Feasibility of the Senhance Surgical System in bariatric surgery | During operation, up to 2 hours
  Conversion rate
Feasibility of the Senhance Surgical System in bariatric surgery | at hospital discharge, up to 30 days
  Length of hospital stay
Feasibility of the Senhance Surgical System in bariatric surgery | up to 30 days postoperatively
  Rehospitalisation rate

CONTACTS AND LOCATIONS:
Overall Officials: Philipp C Nett, MD, Study Director — Inselspital Universitätsspital Bern
Locations (1):
- Inselspital Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-11-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT05208138/Prot_000.pdf